CLINICAL TRIAL: NCT06311292
Title: Pilot Study of Intrapulmonary Percussive Ventilation for Sputum Induction in Adults With Cystic Fibrosis
Brief Title: Intrapulmonary Percussive Ventilation for Sputum Induction in Adults With Cystic Fibrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Daniel J. Weiner (Other)
Responsible Party: Sponsor-Investigator, Daniel J. Weiner, Professor of Pediatrics and Pediatric Pulmonologist, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STUDY22090138
Record Dates: First submitted 2024-03-07; First posted 2024-03-15 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-02

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Masking Description: No parties will be prevented from having knowledge of the Volara System use.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Intrapulmonary Percussive Ventilation for Non-sputum Producer (Experimental): Unable to produce adequate amount of lower airway bacterial sampling for culture results in last year.
  Interventions: Device: Volara System

INTERVENTIONS:
Device: Volara System — Intrapulmonary percussive ventilation for mobilizing mucus.

SUMMARY:
This is a small pilot study with the goal of identifying a superior sputum collection method in Cystic Fibrosis patients unable to produce a sputum.

Participants will use the Volara System during clinic visit in an attempt to produce sputum.

DETAILED DESCRIPTION:
Since the introduction of CFTR modulator therapies, most patients with Cystic Fibrosis (CF) have been unable to produce an adequate sputum sample for clinical monitoring. COVID-19 also presented a safety concern for staff and patients that may become exposed during sputum induction performed in the clinic rooms due to lack of negative pressure rooms and especially for patients who were unvaccinated. These issues led to lack of microbiology data for clinical care.

The purpose of this project is to identify a superior sputum collection method for those patients unable to produce a sputum to guide future antimicrobial management.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years or older
2. 2. Currently prescribed hypertonic saline treatment as part of routine airway clearance therapy.

2. No sputum culture results in last one year or those who were unable to produce sputum from VPEP method used in QI project 3771

Exclusion Criteria:

1. < 18 years old
2. Sputum culture results in last one year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-05-29 (Actual); Primary Completion 2025-03-19 (Actual); Study Completion 2025-03-19 (Actual)

PRIMARY OUTCOMES:
Sufficient sputum quantity for a pellet | 10 minutes
  Percentage of patients with a successful culture result from sputum

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Weiner, MD, Principal Investigator — UPMC Children's Hospital of Pittsburgh
Locations (1):
- UPMC Presbyterian Hospital, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
The investigators do not currently have an individual participant data sharing plan. However, de-identified research data/documents may be shared in the future with other investigators who share similar research interests.
  Specimens and data will not be released without (1) PI written permission and (2) appropriate Institutional Review Board (IRB) approval. Data use and/or material transfer agreements will also be required as applicable to outside researchers.